CLINICAL TRIAL: NCT00789815
Title: Sedation for Flexible Bronchoscopy and Real Time Endobronchial Ultrasound -A Comparison Between Bispectral Index-guided Sedation and Conventional Sedation
Brief Title: Bispectral Index-guided Sedation for Flexible Bronchoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Ting-Yu Lin, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 97-0257B
Record Dates: First submitted 2008-11-10; First posted 2008-11-13 (Estimated); Results first posted 2010-04-20 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2010-04

CONDITIONS: Flexible Bronchoscopy
Keywords: flexible bronchoscopy; sedation; bispectral index

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BIS-guided propofol infusion (Active Comparator): In the study group, induction was started using alfentanil 4~5μg/kg bolus following repeated propofol boluses (0.5~1.5 mg/kg) until the BIS level reached 70. During maintenance, propofol infusion (3~12 mg/kg/hour) was given using a syringe pump (Injectomat Agilia, Fresenius Kabi, France), which was titrated to keep the BIS level between 65 and 75.
  Interventions: Device: Bispectral index guide propofol infusion
- Clinical-judged midazolam administration (Active Comparator): In the control group, induction was started using alfentanil 4~5μg/kg bolus following 2 mg midazolam bolus. After 2 minutes, if the patient was not well sedated, midazolam boluses were repeat by increments of 2 mg/2min until conscious sedation was achieved
  Interventions: Drug: Clinical-judged midazolam administration

INTERVENTIONS:
Device: Bispectral index guide propofol infusion — Induction:
  Alfentanil: 5μg/kg slowly push. Propofol: 0.5-1.5mg/kg slowly push till BIS value 70.
  Maintenance:
  Propofol infusion (3~12 mg/kg/hour) to maintain BIS around 65~75. Alfentanil: 5μg/kg slowly push Q15min prn if severe cough.
  Other Names: BIS-guided profopol infusion
  Arms: BIS-guided propofol infusion
Drug: Clinical-judged midazolam administration — Induction:
  Alfentanil: 5μg/kg slowly push. Midazolam: 2 mg slowly push followed by increments of 2 mg/ 2min till OAA/S* 2~3.
  Maintenance:
  Midazolam: 2 mg/ 2min prn to keep OAA/S* 2~3 or if intolerance of procedure. Alfentanil as study arm.
  *Observer's assessment of alertness/sedation (OAA/S):
  Class 5: Responds readily to name spoken in normal tone.
  Class 4: Lethargic response to name called in normal tone.
  Class 3: Responds only to name called loudly.
  Class 2: Responds only to shaking.
  Class 1: No response to shaking.
  Arms: Clinical-judged midazolam administration

SUMMARY:
With the advances of flexible bronchoscopy, like metallic stent, electrocautery and real time endobronchial ultrasound, the complexity and duration of procedures are increasing. So, adequate sedation and analgesia is important for both patients and bronchoscopist.

Clinical-judged midazolam administration is the current standard. However, midazolam is difficult to titrated and the clinical observations are not reliable sedative indices. Propofol is titrated easily because of its unique pharmacokinetics. Bispectral index (BIS), a real time monitor of depth-of-sedation, has been applied in general anesthesia.

We design a BIS-guided propofol sedation for bronchoscopy. Through the combination of advantages of propofol and BIS, we hope to provide patients a more tolerable and safety sedation for bronchoscopy.

DETAILED DESCRIPTION:
It is well known that patients undergoing bronchoscopy could be less suffering and the procedures could be carried on more smoothly if the patients have adequate sedation and analgesia. The preferred sedative and analgesic drugs are Midazolam and opioid, like Alfentanil or Morphine, which were titrated according to physicians' judgment on patients' clinical responsiveness. However, due to the pharmacokinetic characteristic of midazolam while used in intravenous injection (onset time 4-6 minutes, effective time 2-4 hours), the effective onset time may be too slow for repeated injection while patients already suffered from the bronchoscopic procedure. It is also noted that when over-sedation occurred the side effects like apnea/hypopnea, hypoxemia, and hypotension could last from dozen minutes to few hours. Although events mentioned above could be handled properly under experienced medical staff, it is still very difficult to predict the oncoming events as the pharmacokinetic effect is variant individually. Ideally, it will be more safe and efficient, during invasive procedure like bronchoscope, if the sedative drug could be onset or vanish fast and the drug effect could be titrated with an objective device directly monitoring the depth of sedation or anesthesia.

Propofol is a short-acting intravenous sedative agent used for the induction of general anesthesia for children and adults; maintenance of general anesthesia; and sedation in medical contexts, such as intensive care unit (ICU) sedation for intubated, mechanically ventilated adults, and in procedures such as colonoscopy. Its mechanism of action is uncertain, but it is postulated that its primary effect may be potentiation of the Gamma-Amino Butyric Acid-A receptor, possibly by slowing the channel closing time. It has a fast onset time (1~2 minutes) but a short working duration (8~10 minutes), which vanished fast after stop administration. Bispectral Index (BIS), an non-invasive neurophysiologic monitor instrument, can transform the electroencephalogram (EEG) and electromyography of the patient to a continual numeral, ranging from 0 to 99, which provides a direct and real-time sedative depth monitor. A BIS value of 0 equals EEG silence, near 100 is the expected value in a fully awake adult, and below70 indicated the patient lose explicit memory recall but still has the ability to maintain his own vital signs.

In this study, we design a sedative technique for bronchoscopy, a BIS-guided propofol administration, to compare with the traditional sedative technique, clinical-judged midazolam administration. Through the combination of the advantages of unique pharmacokinetics of propofol and real time monitor of sedative level from BIS, we hope to provide patients undergoing bronchoscopy a more satisfied and safety sedative procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients (>18 years old) requiring elective flexible bronchoscopy or Real time endobronchial ultrasound with transbronchial needle aspiration.

Exclusion Criteria:

* American Society of Anesthesiologists classification of physical status 4 and 5, including hepatic or renal failure, severe obstructive sleep apnea and severe chronic obstructive pulmonary disease.
* Significant Central nervous system disorders or other factors contributing to access consciousness difficultly.
* Allergic history to study drugs.
* A history of glaucoma in the midazolam arm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2008-04; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ting-Yu Lin, MD, Principal Investigator — Division of Thoracic Medicine, Chang Gung Memorial hospital
Locations (1):
- Division of Thoracic Medicine, Chang Gung Memorial Hospital, Taoyuan, Taiwan

REFERENCES:
- [Derived] Lo YL, Lin TY, Fang YF, Wang TY, Chen HC, Chou CL, Chung FT, Kuo CH, Feng PH, Liu CY, Kuo HP. Feasibility of bispectral index-guided propofol infusion for flexible bronchoscopy sedation: a randomized controlled trial. PLoS One. 2011;6(11):e27769. doi: 10.1371/journal.pone.0027769. Epub 2011 Nov 23. PMID 22132138

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The investigator evaluate the inclusion and exclusion criteria of patients undergoing flexible bronchoscopy (FB) at the bronchoscopic room. If patients were eligible, investigator would explain the informed concent, the safety managements and the way of sedation and FB to patients.
Pre-assignment Details: If patients or family refused to join the study later or if the intravenous catheter was difficultly placed on the forearm, patients were excluded before assignment.
Groups:
- Clinical-judged Midazolam Administration: In the control group, induction was started using alfentanil 4~5μg/kg bolus following 2 mg midazolam bolus. After 2 minutes, if the patient was not well sedated, midazolam boluses were repeat by increments of 2 mg/min until conscious sedation was achieved
Period: Overall Study
Arm/Group | BIS-guided Propofol Infusion | Clinical-judged Midazolam Administration
Started | 250 | 250
Completed | 243 | 249
Not Completed | 7 | 1
Not completed — Protocol Violation | 6 | 1
Not completed — Intubation due to massive bleeding | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BIS-guided Propofol Infusion | Clinical-judged Midazolam Administration | Total
Number analyzed (Participants) | 250 | 250 | 500
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 144 | 124 | 268
  >=65 years | 106 | 125 | 231
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (13.1) | 62.0 (14.7) | 60.9 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 111 | 213
  Male | 148 | 139 | 287
Region of Enrollment [Number; unit: participants]
  Taiwan | 250 | 250 | 500

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Any Hypoxemia Event During Flexible Bronchoscopy
Description: The hypoxemia event is defined as that when the oxyhemoglobin (SpO2) was less than 90% with any duration during the flexible bronchoscopy.
Time Frame: From the time when bronchoscope introducing patients' nose or mouth to the time when bronchoscope leaving patients' nose or mouth
Population: Patients completed the whole intervention.
Measure: Number; unit: participants
Arm/Group | BIS-guided Propofol Infusion | Clinical-judged Midazolam Administration
Number analyzed (Participants) | 243 | 249
participants | 97 | 88
Statistical Analysis 1: Comparison: BIS-guided Propofol Infusion vs Clinical-judged Midazolam Administration; The null hypothesis: the incidence of hypoxemia occured during FB with BIS-guided propofol infusion is higher than that with clinical-judged midazolam administration. Power calculation is described below; Test type: Non-Inferiority or Equivalence — A preliminary study was performed to determine the sample size before this trial. 15 and 15 patients undergoing FB received BIS-guided propofol sedation and clinical-judged midazolam sedation, respectively. The incidences of hypoxemia were 0.33 and 0.20, respectively. The selected sample size of 225 in each group will yield 90% power for detecting a clinically meaningful difference of 0.13 at the 5.0% level of significance. To allow for 10% missing data, we recruited 250 patients per group; p = 0.05, Chi-squared

2. Primary Outcome: The Number of Participants With Any Hypotension Event During Flexible Bronchoscopy
Description: The event of hypotension: when the systolic blood pressure (SBP) was less than 90mmHg with any duration.
Time Frame: as for outcome 1
Population: patients completed the whole intervention
Measure: Number; unit: participants
Arm/Group | BIS-guided Propofol Infusion | Clinical-judged Midazolam Administration
Number analyzed (Participants) | 243 | 249
participants | 18 | 11
Statistical Analysis 1: Comparison: BIS-guided Propofol Infusion vs Clinical-judged Midazolam Administration; The null hypothesis: the incidence of hypotension during FB in patients of study group is higher than that in the control group; Test type: Superiority or Other; p = 0.05, Chi-squared

3. Secondary Outcome: The Number of Participants Causing Any Procedure Interference by the Patients' Movement During Flexible Bronchoscocopy
Description: "Procedure interference by patients' movement" was when the bronchoscopist had to stop the procedure temporarily and our assistant had to hold down the irritant patient
Time Frame: as for outcome 1
Measure: Number; unit: participants
Arm/Group | BIS-guided Propofol Infusion | Clinical-judged Midazolam Administration
Number analyzed (Participants) | 243 | 249
participants | 33 | 90
Statistical Analysis 1: Comparison: BIS-guided Propofol Infusion vs Clinical-judged Midazolam Administration; Test type: Superiority or Other; p = 0.05, Chi-squared

4. Secondary Outcome: The Number of Participants Causing Any Procedure Interference by Cough
Description: "Procedure interference by cough" was when the bronchoscopist had to stop the procedure temporarily and additional xylocaine spray and/or alfentanil had to be given to stop the cough.
Time Frame: as for outcome 1
Measure: Number; unit: participants
Arm/Group | BIS-guided Propofol Infusion | Clinical-judged Midazolam Administration
Number analyzed (Participants) | 243 | 249
participants | 73 | 110
Statistical Analysis 1: Comparison: BIS-guided Propofol Infusion vs Clinical-judged Midazolam Administration; Test type: Superiority or Other; p = 0.05, Chi-squared

5. Secondary Outcome: The Recovery Time to Orientation
Description: The time to orientation defined as the time between finishing flexible bronchoscopy to the moment when patients could open their eyes spontaneously, could recall their date of birth, and perform a finger-nose test correctly
Time Frame: After the bronchoscope leaving patients' nose or mouth to the time patients returned orientation
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | BIS-guided Propofol Infusion | Clinical-judged Midazolam Administration
Number analyzed (Participants) | 243 | 249
minutes | 11.7 (10.2) | 30.0 (26.8)
Statistical Analysis 1: Comparison: BIS-guided Propofol Infusion vs Clinical-judged Midazolam Administration; Test type: Superiority or Other; p = 0.05, t-test, 2 sided

6. Primary Outcome: The Global Tolerance for Flexible Bronchoscopy by Verbal Analogus Scale
Description: The global tolerance of the entire procedure was evaluated on a 10-point verbal analogous scale (VAS, 0: no bother, 10: worst intolerable).
Time Frame: After patients recovered orientation and before they leaved the scope room.
Population: Patients received intervention completely
Measure: Median (Full Range); unit: units on a scale
Arm/Group | BIS-guided Propofol Infusion | Clinical-judged Midazolam Administration
Number analyzed (Participants) | 243 | 249
units on a scale | 0 [0 to 10] | 0 [0 to 10]
Statistical Analysis 1: Comparison: BIS-guided Propofol Infusion vs Clinical-judged Midazolam Administration; The null hypothesis: the global tolerance of patients in study is worse than that in the control group; Test type: Superiority or Other; p = 0.05, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: The Recovery Time to Ambulation
Description: The recovery time to ambulation defined as the time between finishing flexible bronchoscopy to the moment when patients could walk without assistance.
Time Frame: After the bronchoscopy
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | BIS-guided Propofol Infusion | Clinical-judged Midazolam Administration
Number analyzed (Participants) | 243 | 249
Minutes | 30.0 (18.2) | 55.7 (40.6)
Statistical Analysis 1: Comparison: BIS-guided Propofol Infusion vs Clinical-judged Midazolam Administration; Test type: Superiority or Other; p = 0.05, t-test, 2 sided

8. Secondary Outcome: Patients Willing Return if Repeated Bronchoscopy is Indicated.
Description: Patients were asked their willingness to return for another FB if needed by means of a five-point scale (definitely not, probably not, unsure, probably would, and definitely would return). Both "probably would", and "definitely would return" were defined as patients agreed to return.
Time Frame: After patients recovered orientation and before they leaved the scope room.
Population: Patients who answered the question in the questionnaire after bronchoscopy
Measure: Number; unit: participants
Arm/Group | BIS-guided Propofol Infusion | Clinical-judged Midazolam Administration
Number analyzed (Participants) | 221 | 226
participants | 171 | 169
Statistical Analysis 1: Comparison: BIS-guided Propofol Infusion vs Clinical-judged Midazolam Administration; Test type: Superiority or Other; p = 0.05, Chi-squared

ADVERSE EVENTS:
Time Frame: During bronchoscopy and after recovery within 3 days.
Description: The adverse events is the primary outcome of this study. So, regular assessment would be done during bronchoscopy and after recovery. In this study, all adverse events recovered spontaneously or after proper managements.
Arm/Group | BIS-guided Propofol Infusion | Clinical-judged Midazolam Administration
Serious Adverse Events (participants affected / at risk) | 2/250 | 0/250
Other Adverse Events (participants affected / at risk) | 115/250 | 100/250
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIS-guided Propofol Infusion (N=250) | Clinical-judged Midazolam Administration (N=250)
Intubation due to massive bleeding after bronchial biopsy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Bleeding from the biopsy site is the risk of bronchial biospy. After intubation, the patient was stabilized. He recovered later and discharged without sequelae.
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Pneumothorax is the risk of transbronchial lung biopsy. After chest tube draining, the patient recovered and discharged without any sequelae.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIS-guided Propofol Infusion (N=250) | Clinical-judged Midazolam Administration (N=250)
Hypoxemia during flexible bronchoscopy (Respiratory, thoracic and mediastinal disorders) | 97 (131) | 89 (131) — The hypoxemia is the risk of bronchoscopy and sedation. This the primary outcome of this study.
Hypotension during flexible bronchoscopy (Cardiac disorders) | 18 (37) | 11 (27) — The hypotension is the risk of sedation. This is the primary outcome of this study.

LIMITATIONS AND CAVEATS:
The bronchoscopists were not blinded to sedative procedures. It was difficult to accomplish totally blind conditions. The bronchoscopist would realize which protocol it was when only observing responses of the investigator.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes